CLINICAL TRIAL: NCT01586312
Title: Treatment of Knee Osteoarthritis With Allogenic Mesenchymal Stem Cells (MSV*) *MSV: Mesenchymal Stromal Cells From Valladolid
Brief Title: Treatment of Knee Osteoarthritis With Allogenic Mesenchymal Stem Cells
Acronym: MSV_allo
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: University of Valladolid (Other); Sanidad de Castilla y León (Other); Centro Medico Teknon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TerCel004; 2011-005321-51 (EudraCT Number); EC11-309 (Other Grant/Funding Number: Spanish Ministry of Health, Independent Clinical Investigatio); MSV_allo (Registry Identifier: Protocol code)
Record Dates: First submitted 2012-04-23; First posted 2012-04-26 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis, Knee; Arthritis of Knee; Knee Osteoarthritis
Keywords: Knee degenerative disease; osteoarthritis; gonarthrosis; stem cell; cellular therapy; regenerative therapy; Mesenchymal stem cells; Bone marrow; musculoskeletal Diseases; Mesenchymal Stromal Cells (allogenic)
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Musculoskeletal Diseases | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allogenic mesenchymal stromal cells injection (Experimental): Mesenchymal stem cells (MSC) prepared from bone marrow from healthy donor expanded ex vivo for 3-4 weeks. Intraarticular injection of 40 millions MSC.
  Interventions: Other: Allogenic mesenchymal stromal cells injection
- Hyaluronic acid (Durolane) (Active Comparator): Intraarticular injection of hyaluronic acid (60 mg)
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Other: Allogenic mesenchymal stromal cells injection — Mesenchymal stem cells prepared from bone marrow of healthy donors and expanded for 3-4 weeks according to our procedure described in PEI Num. 10-134, authorized by the Spanish Medicine Agency
  Other Names: MSV; Mesenchymal Stem Cells; MSC
  Arms: Allogenic mesenchymal stromal cells injection
Drug: Hyaluronic Acid — Intra-articular injection of 60 mg of hyaluronic acid (Durolane) in a single injection (3 ml)
  Other Names: Hyaluronic acid, durolane, CE mark:516407
  Arms: Hyaluronic acid (Durolane)

SUMMARY:
In this study we want to evaluate the clinical use of allogenic mesenchymal stem cells (MSC), obtained from bone marrow of healthy donors, for treatment of knee osteoarthritis. The trial is based in our own previous results with autologous MSC (ongoing NCT01183728 trial). We propose here a multicenter, phase I-II clinical trial, prospective, randomized, blinded, and controlled for the treatment of osteoarthritis (degrees II and III and IV). The assay consists of two arms with 15 patients each one. Patients in the experimental arm will be given an intra-articular transplantation of allogenic MSC, expanded "Ex Vivo" with our GMP-compliant procedure (MSV, PEI No. 10-134, authorized by the Competent Authority; same as in NCT01183728). In the control arm a standard treatment with intra-articular injection of hyaluronic acid shall be given. We shall follow the evolution of pain, disability, quality of life and quantitative changes in structure and composition of cartilage determined by T2-weighted MRI relaxation (Cartigram) for one year.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis grade II, III and IV of Kellgren and Lawrence assessed by two observers.
* Chronic knee pain with mechanical characteristics.
* No local or systemic septic process.
* Haematological and biochemical analysis without significant alterations that contraindicate treatment.
* Informed written consent of the patient.
* The patient is able to understand the nature of the study

Exclusion Criteria:

* Age over 75 or under 18 years or legally dependent
* Present Infection (to be included in the study no signs of infection must be evidenced)
* Congenital or acquired malformation resulting in significant deformity of the knee (varus<10º; valgus<20º) and leading to problems in application or evaluation of results.
* Overweight expressed as body mass index (BMI) greater than 30.5 (obesity grade II). BMI estimated as mass (kg) / corporal surface (m2).
* Women who are pregnant or intend to become pregnant or breast-feeding
* Neoplasia
* Immunosuppressive states
* Intra-articular infiltartion of any treatments in the last 3 months previous to study inclusion
* Participation in another clinical trial or treatment with a different investigational product within 30 days prior to inclusion in the study.
* Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier García-Sancho, MD, PhD, Study Chair — University of Valladolid, Scientific Park; Aurelio Vega, MD,PhD, Study Director — Hospital Clinico Universitario, Valladolid; Luis Orozco, MD, PhD, Study Director — Centro Médico Teknon, Barcelona; Ana Sanchez, MD, PhD, Study Director — Director, Cell Production Unit, Parque Científico UVa; Jose M Moraleda, MD. PhD, Study Director — Virgen de la Arrixaca University Hospital, Murcia, Spain
Locations (2):
- Spain (2):
  - Centro Medico Teknon, Barcelona, Barcelona
  - Hospital Clinico Universitario, Valladolid, Valladolid

REFERENCES:
- [Background] Orozco L, Soler R, Morera C, Alberca M, Sanchez A, Garcia-Sancho J. Intervertebral disc repair by autologous mesenchymal bone marrow cells: a pilot study. Transplantation. 2011 Oct 15;92(7):822-8. doi: 10.1097/TP.0b013e3182298a15. PMID 21792091
- [Background] Orozco L, Munar A, Soler R, Alberca M, Soler F, Huguet M, Sentis J, Sanchez A, Garcia-Sancho J. Treatment of knee osteoarthritis with autologous mesenchymal stem cells: a pilot study. Transplantation. 2013 Jun 27;95(12):1535-41. doi: 10.1097/TP.0b013e318291a2da. PMID 23680930
- [Background] Orozco L, Munar A, Soler R, Alberca M, Soler F, Huguet M, Sentis J, Sanchez A, Garcia-Sancho J. Treatment of knee osteoarthritis with autologous mesenchymal stem cells: two-year follow-up results. Transplantation. 2014 Jun 15;97(11):e66-8. doi: 10.1097/TP.0000000000000167. No abstract available. PMID 24887752
- [Derived] Vega A, Martin-Ferrero MA, Del Canto F, Alberca M, Garcia V, Munar A, Orozco L, Soler R, Fuertes JJ, Huguet M, Sanchez A, Garcia-Sancho J. Treatment of Knee Osteoarthritis With Allogeneic Bone Marrow Mesenchymal Stem Cells: A Randomized Controlled Trial. Transplantation. 2015 Aug;99(8):1681-90. doi: 10.1097/TP.0000000000000678. PMID 25822648
- See also: Cell Therapy Network — http://www.red-tercel.com
- See also: osteoarthritis, knee — http://www.ncbi.nlm.nih.gov/mesh/68020370
- See also: mesenchymal stem cells — http://www.ncbi.nlm.nih.gov/mesh?term=cell%2C%20mesenchymal%20stem

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 patients were included between 26/Jul/2012 (Pat. 01) and12/Dic/2012 (Pat. 30).
Pre-assignment Details: All patients fulfilled the selection criteria, were randomized and received the assigned medication.
Groups:
- Allogenic Mesenchymal Stromal Cells: Mesenchymal stem cells (MSC) prepared from bone marrow from healthy donor expanded ex vivo for 3-4 weeks. Intraarticular injection of 40 millions MSC.
  Injection of Mesenchymal Stromal Cells: Mesenchymal stem cells prepared from bone marrow of healthy donors and expanded for 3-4 weeks according to our procedure described in PEI Num. 10-134, authorized by the Spanish Medicine Agency
Period: Overall Study
Arm/Group | Allogenic Mesenchymal Stromal Cells | Hyaluronic Acid (Durolane)
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allogenic Mesenchymal Stromal Cells | Hyaluronic Acid (Durolane) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.60 (9.57) | 57.33 (9.41) | 56.97 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Adverse events reported. Clinical review and questionaires for pain, disability and quality of life at 0, 3, 6 and 12 months
Time Frame: Up to one year
Population: Efficacy evaluable patients (EEP): A patient has been considered evaluable whenever it has undergone the specified interventions (injection of hyaluronic acid or allogeneic MSC).
  and
  Safety population (SP): The population that includes all evaluable patients who have undergone one of the two study treatments.
Measure: Number; unit: participants
Arm/Group | Allogenic Mesenchymal Stromal Cells | Hyaluronic Acid (Durolane)
Number analyzed (Participants) | 15 | 15
participants | 14 | 13

2. Secondary Outcome: Pain and Disability Evolution (WOMAC, Visual Analogue Scale, Lequesne Index and SF-12 Scores)
Description: Clinical review, questionaires for pain, disability and quality of life at 0, 3, 6 and 12 months.
  WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index): Questionnaire to quantify the pain, stiffness and physical function in patients with osteoarthritis of the knee or hip.
  SF-12 (Short Form 12, an abbreviated form of SF36) is a questionnaire for the detection of changes in quality of life.
  The visual analogue scale (VAS) is a psychometric response scale which can be used for subjective measurements of knee pain.
  LEQUESNE algofunctional index: is a composite measure of pain and disability, with specific self-report questionnaires for knee (osteoarthritis).
  All the scale ranges ranges (minimum and maximum scores) are between 0 and 100%.
  Values are given in differences from baseline (usually negative values). More negative values show more improvement on both scales.
Time Frame: up to one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allogenic Mesenchymal Stromal Cells | Hyaluronic Acid (Durolane)
Number analyzed (Participants) | 15 | 15
units on a scale
  WOMAC11_Changes from Basal - General 3 months | -8.48 (22.6) | -4.52 (17.4)
  WOMAC11_Changes from Basal - General 6 months | -13.03 (18.2) | -5.47 (15.9)
  WOMAC11_Changes from Basal - General 12 months | -13.47 (22.8) | -4.10 (18.4)
  WOMAC11_Changes from Basal - Dificulty 3 months | -8.51 (22.8) | -6.46 (18.7)
  WOMAC11_Changes from Basal - Dificulty 6 months | -14.53 (19.8) | -6.97 (20.5)
  WOMAC11_Changes from Basal - Dificulty 12 months | -12.59 (23.1) | -4.26 (21.3)
  WOMAC11_Changes from Basal - Stiffness 3 months | -4.77 (30.5) | -1.93 (25.2)
  WOMAC11_Changes from Basal - Stiffness 6 months | -3.17 (23.8) | -2.87 (23.6)
  WOMAC11_Changes from Basal - Stiffness 12 months | -10.67 (31.1) | -4.50 (29.5)
  WOMAC11_Changes from Basal - Pain 3 months | -10.01 (23.7) | -4.27 (17.2)
  WOMAC11_Changes from Basal - Pain 6 months | -13.02 (19.0) | -5.97 (12.1)
  WOMAC11_Changes from Basal - Pain 12 months | -16.30 (23) | -6.36 (15.8)
  SF-12_Changes from Basal - General Health 3 months | 0.12 (22.5) | 0.39 (16.2)
  SF-12_Changes from Basal - General Health 6 months | 10.64 (22.8) | 2.11 (21.2)
  SF-12_Changes from Basal - General Health 12 month | 5.24 (27.9) | 2.51 (21.1)
  SF-12_Changes from Basal - Physical function 3 m | 10.00 (36.4) | 18.33 (30.6)
  SF-12_Changes from Basal - Physical function 6 m | 13.33 (26.5) | 11.67 (32.6)
  SF-12_Changes from Basal - Physical function 12 m | 21.67 (22.9) | 20.00 (30.2)
  SF-12_Changes from Basal - Physical rol 3 months | 2.50 (21.2) | 4.17 (31.2)
  SF-12_Changes from Basal - Physical rol 6 months | 6.67 (38.9) | 9.17 (29.7)
  SF-12_Changes from Basal - Physical rol 12 months | 5.00 (34.0) | 6.67 (30.6)
  SF-12_Changes from Basal - Emotional rol 3 months | -1.67 (22.6) | -5.83 (24.5)
  SF-12_Changes from Basal - Emotional rol 6 months | 5.83 (33.0) | 1.67 (15.6)
  SF-12_Changes from Basal - Emotional rol 12 months | 0.00 (31.0) | 0.83 (18.0)
  SF-12_Changes from Basal - Body pain 3 months | 10.0 (26.4) | 5.00 (28.7)
  SF-12_Changes from Basal - Body pain 6 months | 15.00 (28.0) | 11.67 (26.5)
  SF-12_Changes from Basal - Body pain 12 months | 13.33 (36.4) | 13.33 (24.8)
  SF-12_Changes from Basal - Mental Health 3 months | -5.83 (24.5) | 3.33 (19.7)
  SF-12_Changes from Basal - Mental Health 6 months | 3.33 (25.2) | 3.33 (19.7)
  SF-12_Changes from Basal - Mental Health 12 months | 0.00 (14.2) | 5.00 (18.8)
  SF-12_Changes from Basal - Vitality 3 months | -6.67 (37.2) | 1.67 (25.8)
  SF-12_Changes from Basal - Vitality 6 months | -1.67 (33.4) | 1.67 (25.8)
  SF-12_Changes from Basal - Vitality 12 months | -8.33 (36.2) | -6.67 (24.0)
  SF-12_Changes from Basal - Social function 3 mo | -1.67 (27.5) | -1.67 (27.5)
  SF-12_Changes from Basal - Social function 6 mo | 6.67 (27.5) | -6.67 (29.1)
  SF-12_Changes from Basal - Social function 12 mo | 6.67 (29.1) | 0.00 (26.7)
  SF-12_Changes from Basal - Physical Health 3 mo | 3.44 (7.8) | 3.71 (7.6)
  SF-12_Changes from Basal - Physical Health 6 mo | 4.51 (7.0) | 3.76 (9.3)
  SF-12_Changes from Basal - Physical Health 12 mo | 5.42 (9.3) | 4.59 (9.3)
  SF-12_Changes from Basal - Mental Health 3 mo | -3.56 (10.5) | -1.99 (8.9)
  SF-12_Changes from Basal - Mental Health 6 mo | 0.44 (11.7) | -1.09 (7.0)
  SF-12_Changes from Basal - Mental Health 12 mo | -2.41 (8.2) | -1.56 (9.1)
  VAS_Changes from Basal - 3 months | -13.67 (30.7) | -7.53 (23.6)
  VAS_Changes from Basal - 6 months | -20.67 (29.3) | -11.93 (20.6)
  VAS_Changes from Basal - 12 months | -21.20 (28.5) | -13.07 (21.6)
  LEQUESNE_Changes from Basal - 3 months | -3.63 (12.4) | -5.18 (12.8)
  LEQUESNE_Changes from Basal - 6 months | -13.95 (10.8) | -5.46 (13.4)
  LEQUESNE_Changes from Basal - 12 months | -8.76 (12.4) | -3.13 (12.6)

3. Secondary Outcome: Evolution of Cartilage Degeneration by T2 Relaxation Measurements in MRI (Cartigram)
Description: Magnetic Resonance imaging measurements of T2 relaxation (Cartigram) performed at 0, 6 and 12 months to quantify articular cartilage degeneration. The values (in milliseconds) are T1/2 for decay of the T2 MRI signals. Normal values are below 50 ms; values above 50 ms correspond to inflamed cartilage.
  Mean (SD) are expressed as the number of values (of a total of 88 measurements) that are between 50 and 90 ms. A value =<4.4 is considered normal (can be attained by chance). Values above 4.4 are considered pathological. The worst possible is 88.
Time Frame: up to one year
Population: The efficacy endpoint analysis will be based on all patients who have not committed major protocol violations, and have at least one assessment of efficacy of the end graft. 3 patients of the allogenic MSC treatment group were excluded from this analysis because of incomplete measurements.
Measure: Mean (Standard Deviation); unit: number of values (range 0-88)
Arm/Group | Allogenic Mesenchymal Stromal Cells | Hyaluronic Acid (Durolane)
Number analyzed (Participants) | 12 | 15
number of values (range 0-88)
  MRI. Nº of values between 50-90 per visit. 0 | 12.33 (3.5) | 13.53 (5.7)
  MRI. Nº of values between 50-90 per visit. 6 | 9.33 (4.5) | 11.73 (7.5)
  MRI.Nº of values between 50-90 per visit.12. | 8.25 (5.6) | 10.73 (5.5)
  MRI. Change of Nº of measurements. 6 | -3.00 (2.5) | -1.80 (5.8)
  MRI. Change of Nº of measurements.12 | -4.08 (6.0) | -2.80 (4.1)

ADVERSE EVENTS:
Time Frame: 1 year
Description: All patients completed the study successfully. The mean duration of the patients in the study was 12.4 (± 0.6) months, 12.5 (± 0.8) months in the MSV group and 12.4 (± 0.3) months in the hyaluronic acid group.
Arm/Group | Allogenic Mesenchymal Stromal Cells | Hyaluronic Acid (Durolane)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 14/15 | 13/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogenic Mesenchymal Stromal Cells (N=15) | Hyaluronic Acid (Durolane) (N=15)
Artralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 7 (9)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 3 (3) | 2 (3)
Nasofaringitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (2)
Rinitis (Infections and infestations) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dental implant (Surgical and medical procedures) | 0 (0) | 2 (2)
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Amenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Premature menopause (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 2 (12)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Dental pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Leak (General disorders) | 1 (1) | 0 (0)
Artralgia/Artritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Arthralgia/Effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Corneal erosion / Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor must review results communications prior to public release.